CLINICAL TRIAL: NCT05291559
Title: Acceptability and Efficacy of Enterade (VS001) in Children at Risk for Environmental Enteric Dysfunction in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20023567
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Environmental Enteric Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enterade (VS001) (Experimental): 237 mL (8 fluid oz) per os, once daily for 14 days
  Interventions: Dietary Supplement: Enterade
- Placebo (Placebo Comparator): 237 mL (8 fluid oz) per os, once daily for 14 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Enterade — Enterade is a glucose-free, amino acid-based medical food containing specific amino acids (aspartic acid, valine, serine, threonine and tyrosine) in addition to electrolytes and a non-sugar sweetener.
  Other Names: VS001
  Arms: Enterade (VS001)
Dietary Supplement: Placebo — The placebo is an identical product to Enterade except without added amino acids.
  Arms: Placebo

SUMMARY:
This is a pilot study to assess the feasibility and acceptability of a trial of Enterade (VS001) to treat environmental enteric dysfunction in children from a low-income setting. Preliminary data on efficacy will also be obtained.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine tolerability of Enterade (VS001) in stunted Bangladeshi children between 1 and 2 years of age
2. To assess the efficacy of Enterade (VS001) in treatment of environmental enteric dysfunction by comparing improvements in 2-h lactulose mannitol ratio between Enterade (VS001) and a placebo.

Secondary Objectives

1. To assess the adherence to the regimen of 237ml (8 oz) of Enterade daily in children aged 1 to 2 years.
2. To assess Enterade (VS001) efficacy by comparing improvements in fecal measures of intestinal inflammation between Enterade (VS001) and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Length-for-age Z score (LAZ) between -1 and -3 standard deviations
* Lactulose mannitol ratio >0.09

Exclusion Criteria:

* Presence of known congenital or chronic diseases other than malnutrition
* Diarrhea (> 3 unformed stools in a 24-hour window) in the 7 days prior to screening
* Anticipated unavailability for study visits
* A sibling previously enrolled in this study

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Change in appetite | Baseline to 14 days
  Parents will complete a study specific survey which will include questions about child's interest in food and food intake which will yield an appetite score.
Change in gastrointestinal health | Baseline to 14 days
  Parents will complete a study specific survey which will include questions about child's gastrointestinal symptoms such as diarrhea, vomiting, nausea, bloating, or constipation to yield a gastrointestinal health score.
Change in 2 hour Lactulose mannitol ratio | Baseline to 14 days
  Assessment of Lactulose mannitol ratio at baseline and day 14

SECONDARY OUTCOMES:
Residual intervention volume | 14 days
  Summation of daily residual volume of unconsumed study product
Fecal lactoferrin | 14 days
  Assessment of fecal lactoferrin concentration at baseline and day 14
Fecal myeloperoxidase | 14 days
  Assessment of fecal myeloperoxidase concentration at baseline and day 14
Fecal neopterin | 14 days
  Assessment of fecal neopterin concentration at baseline and day 14
Fecal Reg 1 beta | 14 days
  Assessment of fecal Reg 1 beta concentration at baseline and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Donowitz, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No